CLINICAL TRIAL: NCT02776878
Title: A Prospective, Single-arm, Multi-center Clinical Trial Evaluating the Efficacy and Safety of Dasatinib in RefrActory MetAstatic Gastrointestinal Stromal Tumor
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of Dasatinib in Refractory Metastatic GIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Shen Lin, MD，PhD, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRAMA GIST
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental): Dasatinib is given orally 50 mg 2 times a day for the first week, if subject is tolerate, then increased to 70 mg 2 times a day. Dasatinib will be continued until unacceptable toxicity and progression.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib

SUMMARY:
The purpose of this study is to determine whether dasatinib is effective and safe in the treatment of refractory metastatic gastrointestinal stromal tumor

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent/metastatic gastrointestinal stromal tumor (GIST). Immunohistochemically, the detection KIT and/or DOG-1 are/is positive
* Patients must have measurable disease meeting the requirement of RECIST 1.1
* Received the gene mutation detection of c - kit/PDGFRA
* Subjects with mutation in exon 11, in exon 9 and wild type c-kit/PDGFRA have failed to imatinib and sunitinib
* Subjects with primary mutation in exon 17 or 18 have failed to imatinib
* Subjects with primary mutation in exon 11 and secondary mutation in exon 17 or 18 have failed to imatinib
* Subjects with mutation in exon 18 of PDGFRA,have received TKI or not
* Eastern Cooperative Oncology Group (ECOG) performance status = 0-2
* Expected OS ≥3 months
* Ability to understand and the willingness to sign a written informed consent document
* Subject will comply with the study procedures and therapy

Exclusion Criteria:

* Local or metastatic GIST is resectable
* Unable to receive the gene mutation detection of c-kit (c-kitproto-oncogeneprotein)/PDGFRA
* AST and/or ALT > 2.5 times ULN, or Bilirubin >1.5 times upper limit of normal (ULN)
* Neutrophil count < 1.5 x 10^9/L, or Platelet count <75 x 10^9/L, or Hemoglobin<90g/L
* Cr >1.5×ULN
* Other malignancy within the past 5 years except for adequately treated carcinoma in situ of the cervix or cutaneous basal cell carcinoma
* Known brain metastasis, spinal cord compression, carcinomatous meningitis, or cerebral or soft meningeal disease through CT or MRI during screening stage
* Within the past 5 years, subjects have one of the following disease: myocardial infarction, serious/instable angina pectoris, symptomatic congestive heart failure or cerebrovascular accident from coronary/peripheral artery bypass grafting
* Known human immunodeficiency virus positivity
* Joining in other trail
* Women who are pregnant or lactating; No contraception for subject during childbearing period
* Subject with other serious acute and chronic physical or mental problems, or laboratory abnormality, will increase the risks associated with trail or drug. It will also interference the judgment of the results. In the judgment of the investigator, subject is inadequate to participant the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survive, calculated from registration until progression or death | 2 years

SECONDARY OUTCOMES:
Overall survival, overall survival will be calculated from registration until death | 2 years
Adverse drug reactions according to NCI CTCAE v4.0 | 2 years, Tolerability will be assessed based on the frequency and severity of Adverse Drug Reactions (ADR) coded according to NCI CTCAE v4.0.
Objective response, according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria | 2 years
Tumor control probability, defined as CR＋PR＋SD, determined according to RECIST 1.1 criteria | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - No.81 Hospital of Chinese People's Liberation Army, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital , Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided